CLINICAL TRIAL: NCT03279731
Title: Liraglutide 3.0mg/d for the Treatment of Binge Eating Disorder
Brief Title: Binge Eating Liraglutide Intervention
Acronym: BELIEVE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was not meeting recruitment goals.
Sponsor: Kelly Allison (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor-Investigator, Kelly Allison, Associate Professor, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 827450
Record Dates: First submitted 2017-09-06; First posted 2017-09-12 (Actual); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Binge-Eating Disorder
Keywords: eating disorder, pharmacotherapy
MeSH Terms: conditions — Binge-Eating Disorder; Feeding and Eating Disorders | interventions — Liraglutide

STUDY DESIGN:
Intervention Model Description: Single-center, double-blind, randomized placebo-controlled trial with parallel groups.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Novo Nordisk's Clinical Services (CS) will label, package, and ship the labelled study drugs to the Penn's Investigational Drug Service (IDS). Dr. Rockwell from Penn's IDS service will generate the randomization code using a 1:1 randomization scheme of liraglutide and placebo. The first subject to meet the treatment criteria will be assigned the first number in the sequence; each subsequent subject to meet treatment criteria will be assigned the next number in the sequence. Unblinding of the treatment codes will occur after all data have been verified and deemed clean by the data managers and statistician, and right before analysis of the data occurs.
  The code for a particular subject may be broken in a medical emergency if knowing the identity of the treatment allocation would influence the treatment of the subject or if demanded by the subject. Whenever a code is broken, the staff-member breaking the code will record the time, date and reason.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml (Active Comparator): Pre-filled, multi-dose pen that delivers doses of 0.6 mg, 1.2 mg, 1.8 mg, 2.4 mg, or 3 mg via subcutaneous injection. Matching the recommended dosage and administration guidelines of the FDA-approved labeling for the use of liraglutide (Saxenda), the medication will be initiated at 0.6 mg daily for 1 week, and then increased by 0.6 mg/day in weekly intervals until a dose of 3.0 mg/day is achieved. Liraglutide is a glucagon-like peptide-1 (GLP-1) receptor agonist.
  Interventions: Drug: Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml
- Placebo (Placebo Comparator): Pre-filled, multi-dose pen that delivers doses of 0.6 mg, 1.2 mg, 1.8 mg, 2.4 mg, or 3 mg of placebo via subcutaneous injection. The placebo will be initiated at 0.6 mg daily for 1 week, and then increased by 0.6 mg/day in weekly intervals until a dose of 3.0 mg/day is achieved.The inactive ingredients include: disodium phosphate dihydrate, 1.42 mg; propylene glycol, 14 mg; phenol, 5.5 mg; and water for injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml — subcutaneous injection, pre-filled, multi-dose pen that delivers doses of 0.6 mg, 1.2 mg, 1.8 mg, 2.4 mg, or 3 mg (6 mg/mL, 3 mL). Matching the recommended dosage and administration guidelines of the FDA-approved labeling for the use of liraglutide (Saxenda), the medication will be initiated at 0.6 mg daily for 1 week, and then increased by 0.6 mg/day in weekly intervals until a dose of 3.0 mg/day is achieved.
  Arms: Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml
Drug: Placebo — subcutaneous injection, pre-filled, multi-dose pen that delivers doses of 0.6 mg, 1.2 mg, 1.8 mg, 2.4 mg, or 3 mg (6 mg/mL, 3 mL). It is designed to be identical to the pen used for liraglutide (Saxenda). Placebo product inactive ingredients: disodium phosphate dihydrate, 1.42 mg; propylene glycol, 14 mg; phenol, 5.5 mg; and water for injection
  Arms: Placebo

SUMMARY:
The study is a 17-week, single-center, double-blind, parallel-group, randomized placebo controlled trial that will test the efficacy of liraglutide 3.0 mg/d as compared to placebo in reducing the number of binge episodes per week, achieving remission from binge episodes, and in changes in body weight, global BED symptom improvement, cognitive restraint of food intake, dietary disinhibition, perceived hunger, quality of life, and depressed mood at treatment end.

DETAILED DESCRIPTION:
All applicants will be initially screened by phone and/or electronically to determine whether they potentially meet eligibility criteria. Those who appear to meet eligibility criteria and remain interested in the trial will be scheduled for an in-person interview.

The in-person interview will be conducted by a psychologist or Masters' level staff member, who will obtain informed consent and evaluate subjects' behavioral eligibility (i.e., willingness and appropriateness to participate) using structured and semi-structured clinical interviews including: an examination of the applicants' BED symptoms, their mood, suicidality, and other general psychopathology. Participants will also be asked to complete questionnaires assessing eating behavior, demographic characteristics, frequency of specific eating behaviors related to loss of control, risk of substance dependence with the consumption of high fat/sugar foods, alexithymia, night eating syndrome, sleep patterns and quality, and attitudes towards food cravings.

Subjects who remain interested and pass this portion of the assessment will proceed to meet with the study physician or nurse practitioner, who will obtain a medical history and conduct a physical examination to determine medical eligibility. Subjects will also have an electrocardiogram (EKG), fasting blood test, and a urine pregnancy test (for females of child bearing age) to confirm eligibility.

Upon successful completion of the screening visit, subjects will be asked to eat as they normally would for 2 weeks. Once per week over these two weeks they will receive a brief survey through REDcap to assess their binge eating episodes for eligibility.

Subjects who continue to meet eligibility criteria assessed at the screening visit and during the run-in period will be scheduled for a randomization visit at the Center within 3 weeks of their screening.

Subjects will be randomly assigned to the two interventions in equal numbers (i.e., 1:1 ratio). The subject's weight, blood pressure, and pulse will then be measured. Following randomization, all subjects will have a medical visit with the study physician or nurse practitioner who will instruct them in the use of liraglutide 3.0 (as described later) and provide the first month's supply of medication.

After randomization, subjects will return at week 1 to assess rate of response. Subjects will return for study visits every two weeks thereafter, at weeks 3, 5, 7, 9, 11, 13, 15, and 17.

These study visits include a brief medical visit (10-15 minutes) with a physician or nurse practitioner to monitor their response to the medication or any changes in health. Vitals and weight will be taken. Additionally, binge episodes, mood, suicidality, and symptom improvement will be assessed by the psychologist or Masters' level trained study staff. Participants will be asked also to complete questionnaires assessing quality of life, obsessions related to food, and food cravings prior to each treatment visit for the secondary outcomes:

In summary, study visits will consist of the medical visit, completion of written surveys, review of structured interviews with the study staff and review of medication adverse events. These visits are expected to last about 30-40 minutes. The study assessments at week 17 will consist of the previously listed procedures and measures in addition to the questionnaires and blood tests conducted at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. BMI > 30 kg/m2 or BMI ≥ 27 - 29.9 kg/m² in the presence of at least one weight-related comorbid condition, such as binge eating disorder, hypertension, or dyslipidemia. There is no upper BMI limit for this trial.
2. Age ≥ 21 years and ≤ 70 years
3. Meet full DSM 5 criteria for BED

   1. Recurrent episodes of binge eating characterized by both consuming an abnormally large amount of food in a short period of time compared with what others might eat in the same amount of time under the same or similar circumstances and experiencing a loss of control over eating during the episode.
   2. These episodes feature at least 3 of the following:

   i. consuming food more rapidly than normal; ii. eating until uncomfortably full; iii. consuming large amounts of food when not hungry; iv. consuming food alone due to embarrassment; v. feeling disgusted, depressed, or guilty after eating a large amount of food. c. Significant distress about the binge episodes is present. d. Binge episodes must occur, on average, at least once per week for 3 months.
4. All races and ethnicities are included
5. Eligible female subjects will be:

   * non-pregnant, evidenced by a negative urine dipstick pregnancy test
   * non-lactating
   * surgically sterile or postmenopausal, or they will agree to continue to use an accepted method of birth control during the study
6. Ability to provide informed consent before any trial-related activities
7. Subjects must:

   * have a primary care provider (PCP) who is responsible for providing routine care
   * have reliable telephone or Internet service to communicate with study staff
   * understand and be willing to comply with all study-related procedures and agree to participate in the study by giving written informed consent
   * plan to remain in the Philadelphia area for the next 6 months or more

Exclusion Criteria:

1. Pregnant or nursing, or plans to become pregnant in the next 6 months, or not using adequate contraceptive measures
2. Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia syndrome type 2
3. Uncontrolled hypertension (systolic blood pressure ≥ 160 mm Hg or diastolic blood pressure ≥ 100 mm Hg)
4. Type 1 diabetes
5. Type 2 diabetes
6. A combination of fasting glucose ≥ 126 mg/dl, combined with an HbA1c >6.5, will be used to indicate the presence of diabetes, an exclusion criterion
7. Recent history of cardiovascular disease (e.g., myocardial infarction or stroke within the past 6 months), congestive heart failure, or heart block greater than first degree
8. Clinically significant hepatic or renal disease
9. Thyroid disease, not controlled
10. History of malignancy (except for non-melanoma skin cancer) in past 5 years
11. The presence of current anorexia nervosa or bulimia nervosa
12. Current major depressive episode, active suicidal ideation, or lifetime history of suicide attempts. We will exclude participants who have a Patient Health Questionnaire-9 (PHQ-9) [31] score > 15, or a score of > 1 on the suicidal ideation item, as well as any risk of suicidality as measured by a score of 4 or 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS)[32].
13. Psychiatric hospitalization within the past 6 months
14. Self-reported alcohol or substance abuse within the past 12 months, including at-risk drinking (current consumption of ≥ 14 alcoholic drinks per week)
15. Diagnosis current or past psychosis
16. Use in past 3 months of medications known to treat BED (such as lisdexamfetamine), induce significant weight loss (i.e., prescription weight loss medications), or induce weight gain (e.g., chronic use of oral steroids, second generation antipsychotics)
17. Currently receiving behavioral or pharmacological treatment for BED
18. Loss of ≥ 10 lb of body weight within the past 3 months
19. Known or suspected allergy to trial medication(s), excipients, or related products
20. Hypersensitivity to liraglutide or any product components
21. The receipt of any investigational drug within 6 months prior to this trial
22. Previous participation in this trial (e.g., randomized and failed to participate)
23. History of pancreatitis
24. History of gastrointestinal surgery (unless it was an adjustable gastric band that has been removed).

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-09-29 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly C Allison, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennyslvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at university based medical school clinic setting. The first participant was randomized on September 29, 2017; the last participant completed participation on September 6, 2019.
  Note: 9 participants were censored from the trial due to an error in medication/placebo assignment by the Investigational Drug Service. As such, these 9 participants were not considered in any of the analyses presented, leaving 13 in the liraglutide and 14 in the placebo group.
Pre-assignment Details: Participants underwent a 2 week run in to assure that they continued to have binge episodes before being randomized to placebo or liraglutide 3.0 mg.
Period: Overall Study
Arm/Group | Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml | Placebo
Started | 19 | 17
Completed | 13 | 14
Not Completed | 6 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml | Placebo | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.4 (7.9) | 42.1 (12.7) | 44.2 (10.6)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male at birth | 7 | 3 | 10
  Female at birth | 6 | 11 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 14 | 27
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 8 | 8 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27
objective binge episodes per week [Mean (Standard Deviation); unit: binge episodes/week] | 4.90 (0.69) | 2.80 (0.67) | 3.30 (2.13)

OUTCOME MEASURES:

1. Primary Outcome: Binge Episodes
Description: Change in objective binge episodes per week from randomization (week 0) to study end (week 17)
Time Frame: baseline and 17 weeks (or last observation carried forward)
Measure: Mean (Standard Deviation); unit: objective binge episodes per week
Groups:
- Liraglutide: Participants randomized to liraglutide 3.0 mg/d
- Placebo: Participants randomized to placebo
Arm/Group | Liraglutide | Placebo
Number analyzed (Participants) | 13 | 14
objective binge episodes per week | -3.97 (0.56) | -2.50 (.053)

2. Secondary Outcome: Remission From Binge-eating
Description: the percentage of participants (completers) who have achieved remission from binge-eating (no binge episodes between weeks 13 - 17)
Time Frame: 13 to 17 weeks
Population: Remission was calculated for completers who had data from weeks 13-17
Measure: Count of Participants; unit: Participants
Arm/Group | Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml | Placebo
Number analyzed (Participants) | 7 | 8
Participants | 3 | 4

3. Secondary Outcome: Assessment of Improvement of Binge Eating Symptoms
Description: week 17 rating on the interviewer-based Clinical Global Impression of Improvement (CGII) Scale for global assessment of BED symptoms The CGII includes the following rating scale: Compared to the patient's condition at baseline to the project [prior to medication initiation], this patient's condition is: 1 very much improved; 2 much improved; 3 improved; 4 no change; 5 worse; 6 much worse; 7 very much worse.
Time Frame: week 17 (or last observation carried forward)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml | Placebo
Number analyzed (Participants) | 13 | 14
units on a scale | 1.52 (.27) | 1.93 (.26)

4. Secondary Outcome: Change in Body Weight
Description: changes in body weight
Time Frame: baseline and 17 weeks (or last observation carried forward)
Population: Last Observation Carried Forward
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml | Placebo
Number analyzed (Participants) | 13 | 14
kg | -4.7 (0.83) | -0.94 (0.73)

ADVERSE EVENTS:
Time Frame: from the beginning to the end of the 17 week trial
Description: Adverse event data collection occurred at each study visit.
Arm/Group | Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 2/19 | 1/17
Other Adverse Events (participants affected / at risk) | 17/19 | 11/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml (N=19) | Placebo (N=17)
Hospitalization due to vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — Participant notified study staff that he was hospitalized for vomiting . Patient did not want to continue the phone conversation and no other information has been gathered.
laparoscopic cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0) — abdominal pain, nausea and cholecystectomy
Ulcerative colitis flare (Gastrointestinal disorders) | 0 (0) | 1 (1) — Hospitalized from 1/3/18-1/5/18. Treated with Remicade infusion. Reported feeling back to baseline on 1/7/18.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liraglutide (Saxenda) 6Mg/Ml Inj Pen 3Ml (N=19) | Placebo (N=17)
nausea (Gastrointestinal disorders) | 5 (7) | 3 (3)
diarrhea (Gastrointestinal disorders) | 5 (5) | 0 (0)
dry mouth (General disorders) | 3 (3) | 0 (0)
upper respiratory infection (Infections and infestations) | 2 (2) | 1 (1)
indigestion (Gastrointestinal disorders) | 2 (2) | 2 (2)
tachycardua (Cardiac disorders) | 3 (3) | 0 (0)
suicidal ideation (Psychiatric disorders) | 1 (2) | 1 (1)
fatigue (General disorders) | 0 (0) | 1 (1)
depressive symptoms (Psychiatric disorders) | 0 (0) | 1 (1)
gastroenteritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
joint pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
UTI (Renal and urinary disorders) | 0 (0) | 1 (1)
constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
bilateral otitis media (Ear and labyrinth disorders) | 1 (1) | 0 (0)
strep throat (Infections and infestations) | 0 (0) | 1 (1)
flu (Infections and infestations) | 1 (1) | 0 (0)
sty (Eye disorders) | 0 (0) | 1 (1)
cholitis flare (Gastrointestinal disorders) | 0 (0) | 1 (1)
insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
headache (General disorders) | 1 (1) | 0 (0)
vaginal bleeding (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
allergic rhinitis (General disorders) | 0 (0) | 1 (1)
common cold (Infections and infestations) | 0 (0) | 1 (1)
toothache (General disorders) | 0 (0) | 1 (1)
worsening edema (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Error by Investigational Drug Service - randomization key interpreted incorrectly at n=21 n= 6 had 2+ consecutive boxes of same agent and were retained in analyses (data censored after first switch); 6 received same agent consistently; n=9 censored

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT03279731/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT03279731/ICF_001.pdf